CLINICAL TRIAL: NCT02172703
Title: Validation of Non-invasive Absolute Intracranial Pressure Monitoring in Patients After Traumatic Brain Injury and Subarachnoid Hemorrhage
Brief Title: Non-invasive Brain Pressure Monitoring After Trauma or Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier Fandino, MD (Other)
Collaborators: Kaunas University of Technology (Other)
Responsible Party: Sponsor-Investigator, Javier Fandino, MD, Chairman, Department of Neurosurgery, Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: aICP_CH_TBI_SAH
Record Dates: First submitted 2014-06-10; First posted 2014-06-24 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Traumatic Brain Injury (TBI); Subarachnoid Hemorrhage (SAH)
Keywords: TBI; SAH; ICP; non invasive measurement
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-invasive ICP measurement (Other): non-invasive ICP measurement with NON-INVASIVE ICP ABSOLUTE VALUE METER (carried out simultainusly with standard invasive ICP measurement catheter and probes)
  Interventions: Device: Non-invasive ICP measurement device

INTERVENTIONS:
Device: Non-invasive ICP measurement device — The non-invasive ICP measurement device used in this study has been developed in the Telematic Science Laboratory at the Kaunas University of Technology, Lithuania.
  The non-invasive method is based on two-depth TCD technique for simultaneously measuring flow velocities in the intracranial and extracranial segments of the ophthalmic artery (OA).
  Other Names: NON-INVASIVE ICP ABSOLUTE VALUE METER; (Vittamed 205)

SUMMARY:
Introduction: Increased intracranial pressure (ICP) is considered to be the most important intracranial mechanism causing secondary injury in patients admitted after acute traumatic brain injury (TBI) and intracranial haemorrhage (ICB) including subarachnoid haemorrhage (SAH). Currently, ICP can be measured and monitored only using invasive techniques. The two ICP measurement methods available - intraventricular and intraparenchymal - require both a neurosurgical procedure in order to implant the catheter and probes within the brain. The invasiveness of current methods for ICP measurement limits the diagnoses reliability of many neurological conditions in which intracranial hypertension is a treatable adverse event. A reliable, accurate and precise non-invasive method to measure ICP would be of considerable clinical value, enabling ICP measurement without the need of a surgical intervention.

Aim:

The aim of this study is to validate a novel non-invasive ICP measurement device by comparing its measurement with the "gold standard" invasive ICP-measurement by intracranial probe. The device used in this study has been been developed in the Telematic Science Laboratory at the Kaunas University of Technology, Lithuania.

Methods:

The non-invasive ICP measurement method will be assessed prospectively using repeatable simultaneous non-invasive and invasive (standard with intracranial probe) ICP measurements on patients presenting with TBI and SAH. The device method is based on two-depth transcranial doppler (TCD) technique for simultaneously measuring flow velocities in the intracranial and extracranial segments of the ophthalmic artery (OA). The intracranial segment of the OA is compressed by ICP and the extracranial segment of the OA is compressed by the pressure Pe externally applied by the device. Two-depth TCD device is used as an accurate indicator of the balance point (Pe = ICP) when the measured parameters of blood flow velocity waveforms in the intracranial and extracranial segments of OA are identical. The device has the same ultrasound transmission parameters as existing TCD devices and meets all patient safety criteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age ≥ 18 years, admitted after TBI or SAH at the Neurosurgical Department, Kantonsspital Aarau, Switzerland.
* Patients under sedation and ICP monitoring
* Informed consent will be obtained from the relatives prior to initiation of the measurements.
* study inclusion/informed consent from relatives possible between hour 24 to 72 after admission to the hospital

Exclusion Criteria:

* Age < 18 years at study entry.
* Patients with wounds, scars including the front orbital region.
* Perforating or penetrating mechanism of TBI
* Patients with orbital injury or abnormal blood flow in both Ophthalmic Arteries
* Patients with previous retina surgery
* Patients with previous cataract surgery
* Patients with any known ocular condition that may be worsened by sustained eye pressure in the opinion of the subject's ophthalmologist
* Patients with radiological signs of calcification or atheromatose plaques in the internal carotid artery detected by CT or angiography (performed prior and independently of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Simultaneously measured non-invasive and invasive ICP values in mmHg (millimeters of mercury) | Max. 3 times/day - approx. 24hours to 30 days after addmission (as long as patient is monitored with invasive ICPprobe)
  Physiological parameters of TBI or SAH patients of primary interest are simultaneously measured paired non-invasive and invasive ICP values.
  New measurement is only initiated if ICP changes for more than 4mmHg in comparison to proceeding measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Fandino, M.D., Principal Investigator — Department of Neurosurgery, Kantonsspital Aarau, Aarau, Switzerland
Locations (1):
- Kantonsspital Aarau, Department of Neurosurgery, Aarau, Canton of Aargau, Switzerland